CLINICAL TRIAL: NCT01185249
Title: Time of Day and Accurate Weights for Patients With Congestive Heart Failure (CHF)
Brief Title: Congestive Heart Failure Weight Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central DuPage Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-010
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-06

CONDITIONS: Congestive Heart Failure
Keywords: CHF; congestive heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Body weight taken in a standing position (Experimental): Subjects will be weighed in the early morning, as standard of care dictates. They will also be weighed after evening medications are given, around 9pm. The evening weight is not standard, therefore considered the study intervention.
  Interventions: Procedure: Weigh subjects on a scale in the standing position

INTERVENTIONS:
Procedure: Weigh subjects on a scale in the standing position — Subjects will stand on a scale in the mornings, and the evenings for 3 days while hospitalized.

SUMMARY:
Early morning weights to monitor CHF patient's fluid status is common practice but there is a lack of evidence that this is the best practice. The purpose of this study is to determine if there is a difference in net weight gain or loss for hospitalized patients with CHF who are weighed in the evening instead of early morning.

DETAILED DESCRIPTION:
This is a quasi-experimental pilot study with prospective cohort design. Study subjects will be weighed in the early morning and then again in the evening for a minimum of three days. Analysis will be accomplished on data by analysis within-subjects data utilizing the paired t test. Other data to be collected includes dates of hospitalization, demographics, dose and timing of medications, lab results and documentation of comorbid conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* Admitted to hospital with a primary diagnosis of heart failure or fluid overload
* Ambulatory with a medical order to be out of bed
* Able to stand on a scale
* Have no problems with balance

Exclusion Criteria:

* Patients with a primary diagnosis other than heart failure or fluid overload
* Patients diagnosed with renal failure
* Non-English speaking
* Unable to follow directions or consent due to cognitive impairment
* Medical order for bed rest
* Involved in another study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice M Siehoff, DNP, RN-BC, Principal Investigator — Central DuPage Hospital
Locations (1):
- Central DuPage Hospital, Winfield, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Once all admission procedures were completed in the cardiac intermediate unit, the nursing staff asked CHF patients in their care, if they had interest in hearing more about the study. After a verbal "yes", the PI or key personnel met with the patient to explain the study, review the consent form, and after ample time, obtain written consent.
Period: Overall Study
Arm/Group | Body Weight Taken in a Standing Position
Started | 66 (Total number of patients consented to participate.)
Completed | 24 (Data was analyzed for patients with three consecutive days of data.)
Not Completed | 42
Not completed — Patients discharged or change in status | 42

BASELINE CHARACTERISTICS:
Arm/Group | Body Weight Taken in a Standing Position
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (2.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 38
Region of Enrollment [Number; unit: participants]
  United States | 66
Body Weight [Mean (Standard Deviation); unit: kilograms] — Body weight on admission
  kilograms | 85.9 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: The Measurement of the Difference Between Early Morning and Evening Weights for CHF Patients
Time Frame: Mean differences in the morning (5am) weights compared for three consecutive days. Day 1, Day 2, Day 3. Mean difference in the morning (5am) and evening (8pm) weights for three consecutive days. Day 1, Day 2, Day 3.
Population: Patients with three consecutive days of morning and evening weights.
Measure: Mean (Standard Deviation); unit: kilograms
Groups:
- Evening Weights: Patients with both morning and evening weights
- Morning Weight: Weight of study patients in kilograms first thing in the morning.
Arm/Group | Evening Weights | Morning Weight
Number analyzed (Participants) | 29 | 29
kilograms | 2.47 (1.80) | 3.09 (2.06)
Statistical Analysis 1: Comparison: Evening Weights vs Morning Weight; Analysis of within subjects design morning and evening weights. Null hypothesis is that there is no difference between morning and evening weights; Test type: Non-Inferiority or Equivalence — Null hypothesis-no difference in morning and evening weights on three consecutive days; p < .001, t-test, 1 sided; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.51306 to 1.73806], Standard Deviation 3.09
Statistical Analysis 2: Comparison: Evening Weights vs Morning Weight; Test type: Superiority or Other; p = 0.01, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Body Weight Taken in a Standing Position
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 0/66

LIMITATIONS AND CAVEATS:
Pilot study with small sample size in one patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No